CLINICAL TRIAL: NCT07148505
Title: Assessment of Real-world Outcomes Among Patients Treated With Kisqali (Ribociclib)
Brief Title: A Study of Real-world Outcomes Among Patients Treated With Ribociclib
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AUS73
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Hormone receptor-positive; Human epidermal growth factor receptor-2 negative; CDK4/6i; Real-world; Adverse Events
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Ribociclib Cohort: Adult patients with mBC who received 1L treatment with ribociclib in combination with endocrine therapy (ET).
- Ribociclib Cohort: 65+ Years Age Group: Patients aged 65 years or older with mBC who received 1L treatment with ribociclib in combination with ET.
- Ribociclib Cohort: 75+ Years Age Group: Patients aged 75 years or older with mBC who received 1L treatment with ribociclib in combination with ET.

SUMMARY:
The main aim of the study was to evaluate the real-world tolerability and safety of ribociclib as a first-line (1L) treatment among adults with hormone receptor-positive/human epidermal growth factor receptor-2 negative (HR+/HER2-) metastatic breast cancer (mBC).

This study used data from the Flatiron Health Research Database (FHRD). The FHRD is a longitudinal database derived from electronic health records (EHRs) and other real-world data (RWD) sources from cancer care providers across the United States. The dataset generated for this study included de-identified patient-level data for eligible individuals between 1 January 2015 up to the data cutoff date, 30 November 2022.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with mBC on or after 1 January 2015.
* Had HR+/HER2- test results.
* Received ribociclib and endocrine therapy in 1L treatment.
* Patients had a gap of 90 days or less between mBC diagnosis date and the first structured EHR activity (e.g., lab tests and prescriptions) after metastatic diagnosis date.

Exclusion criteria:

None identified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a restrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Number of Patients by Type of Real-world Adverse Event (AE) of Interest During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Real-world AE of Interest at Baseline | Baseline
Number of Patients by Type of Real-world AE of Interest During 1L Treatment Among Those Without the Specific Real-world AE at Baseline | Up to approximately 5 years and 5 months

SECONDARY OUTCOMES:
Number of Patients by Demographic Category | Baseline
  Demographics included:
  * Age at start of 1L treatment (18-64, 65 years or older)
  * Gender
  * Race
  * Ethnicity
Number of Patients by Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * Type of medical practice (academic, community or both)
  * Geographic region
  * Type of health plan
  * Stage of cancer at initial diagnosis
  * Year of metastatic cancer diagnosis
  * Eastern Cooperative Oncology Group (ECOG) performance score
  * Received chemotherapy prior to ribociclib treatment initiation
  * Menopausal status
  ECOG performance score measures a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. Scores range from 0 (fully active, able to carry out all pre-disease performance without restriction) to 5 (deceased).
Clinical Characteristic: Body Mass Index (BMI) | Baseline
Clinical Characteristic: Time Between Initial Diagnosis and Metastatic Diagnosis | Baseline
Clinical Characteristic: Time Between Metastatic Diagnosis and Initiation of 1L Treatment | Baseline
Clinical Characteristic: Duration of Follow-up | Up to approximately 5 years and 5 months
Clinical Characteristic: Number of Patients by Patient Disposition at Data Cutoff | Up to approximately 5 years and 5 months
  Patient disposition included patients who died and discontinued treatment early.
Number of Patients by Year of Treatment Initiation for Each Line of Treatment | Up to approximately 5 years and 5 months
  Lines of treatment included 1L, second-line (2L), and third-line (3L).
Duration of Each Line of Treatment | Up to approximately 5 years and 5 months
  Lines of treatment included 1L, 2L, and 3L.
Number of Patients Still on 1L Treatment at Last EHR Activity | Up to approximately 5 years and 5 months
Number of Patients Still on 2L Treatment at Last EHR Activity | Up to approximately 5 years and 5 months
Number of Patients Still on 3L Treatment at Last EHR Activity | Up to approximately 5 years and 5 months
Number of Patients by Type of ET Partner During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Treatment Category During Each Line of Treatment | Up to approximately 5 years and 5 months
  Lines of treatment included 1L, 2L, and 3L.
  Treatment categories included:
  * Cyclin dependent kinase 4/6 (CDK4/6) inhibitor based regimen
  * Chemotherapy based regimen
  * Clinical study drug
  * ET monotherapy
  * mTor based regimen
  * PI3K based regimen
Number of Patients by Type of CDK4/6 Inhibitor Based Treatment During Each Line of Treatment | Up to approximately 5 years and 5 months
  Lines of treatment included 1L, 2L, and 3L.
  CDK4/6 inhibitor-based treatments included:
  * Ribociclib
  * Abemaciclib
  * Palbociclib
Number of Patients by Total Number of Ribocicilib Dose Reduction Episodes During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Ribociclib Dose at Each Dose Reduction Episode During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Ribociclib Dosing Schedule at Each Dose Reduction Episode During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Status of Oral Therapy at the End of Each Dose Reduction Episode During 1L Treatment | Up to approximately 5 years and 5 months
  Status included continuing, discontinued, dose change, held, not documented, and unknown, patient sent to hospice.
Number of Patients by Reason for Change in Ribociclib Dose During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Reason for Stopping Ribociclib 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Type of Real-world Adverse Event (AE) During 1L Treatment | Up to approximately 5 years and 5 months
Number of Patients by Action Following or in Response to Real-world AE During 1L Treatment | Up to approximately 5 years and 5 months
  Actions included:
  * Hospitalization
  * Treatment for AE
  * Therapy discontinuation
  * Therapy dose or schedule change
  * Therapy hold

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States